CLINICAL TRIAL: NCT06085690
Title: A Multicenter Clinical Translational Study of "ICU-NO CRBSI" Based on Improvement Science in China
Brief Title: Multicenter Clinical Translational Study of "ICU-NO CRBSI" Based on Improvement Science
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Fudan University Evidence-based Nursing Center (Unknown); Shanghai Zhongshan Hospital (Other); Children's Hospital of Fudan University (Other); Shanghai Public Health Clinical Center (Other Government); Shandong First Medical University affiliated Provincial Hospital (Unknown); Affiliated Hospital of Nantong University (Other); Hospital of Obstetrics and Gynecology affiliated to Fudan University (Unknown); Shengjing Hospital (Other); The First Affiliated Hospital of University of South China (Other); East China Hospital Affiliated to Fudan University (Unknown); The First Affiliated Hospital of Dali University (Unknown); Xinjiang Bayingoleng Mongolian Autonomous Prefecture People's Hospital (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Chinese Academy of Medical Sciences (Other); Shanghai Minhang Central Hospital (Other); Xi 'an children's hospital (Unknown); Huashan Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Affiliated Hospital of Guizhou Medical University (Unknown); Affiliated Hospital of Southwest Medical University (Other); Shenzhen Third People's Hospital (Other); Shanghai Dongfang Hospital (Unknown)
Responsible Party: Principal Investigator, ChunLei Li, graduate student, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: B2023-212R
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: CRBSI - Catheter Related Bloodstream Infection; Evidence-based Nursing Practice; Central Venous Catheter Related Bloodstream Infection; Central Venous Catheter Associated Bloodstream Infection; Central Line Infection; CLABSI - Central Line Associated Bloodstream Infection; Quality Improvement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Hospitals were divided into different groups, and the subjects and effect evaluators were blinded because they could not hide the assignment and the implementers were blinded. The main outcome indicators were laboratory objective indicators of CRBSI diagnosis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Existing central venous catheters in the hospital or ICU maintain routine care procedures (No Intervention): According to the hospital or ICU catheterization, maintenance and removal of central venous catheter routine care
- evidence-based intervention Plan for the Prevention of CRBSI in ICU patients (Experimental): On the basis of routine nursing, the "evidence-based intervention Plan for the Prevention of CRBSI in ICU patients" was implemented for intervention.
  Interventions: Behavioral: evidence-based intervention Plan for the Prevention of CRBSI in ICU patients

INTERVENTIONS:
Behavioral: evidence-based intervention Plan for the Prevention of CRBSI in ICU patients — On the basis of routine nursing, the "evidence-based intervention Plan for the Prevention of CRBSI in ICU patients" was implemented for intervention.
  Arms: evidence-based intervention Plan for the Prevention of CRBSI in ICU patients

SUMMARY:
The goal of this type of study is to construct the continuous quality promotion project "ICU-NO CRBSI(Catheter-Related Bloodstream Infection , CRBSI)" based on improvement science, and to verify its effect in the prevention of central venous catheter-related bloodstream infection and continuous quality improvement in ICU ( Intensive Care Unit , ICU) through multi-center implementation and two rounds of improvement.

The main question[s] it aims to answer are:

What is the incidence of catheter-related bloodstream infection in the ICU of participating units? How compliant are health care providers in the ICU with evidence-based sensory control practices for the prevention of catheter-associated bloodstream infection?

Participants will be provided with the hospital's routine CVC (Central Venous Catheter ,CVC) care practices and CVC quality improvement measures based on evidence-based guidelines What technical and cultural support is needed to implement quality and safety improvement measures?

DETAILED DESCRIPTION:
A multicenter, cluster-randomized controlled trial was conducted to verify the effect of the intervention scheme and the improvement strategy.

A continuous sample was taken based on subjects that met the inclusion criteria. This study was a multicenter cluster randomized controlled trial involving 23 research centers/medical institutions, including the Evidence-Based Nursing Center of Fudan University and Zhongshan Hospital affiliated to Fudan University. Co-led by the Pediatric Hospital Affiliated to Fudan University, a total of 23,000 catheter days (about 8050 people) were included, and each center planned to include 1,000 catheter days (about 350 people). Patients admitted to ICU from October to December 2023 were taken as baseline study objects, and ICU patients from January to March 2024 were entered into the control phase of the study experiment. ICU patients from April 2024 to June 2024 were included in the continuous observation group, and from July 2024 to September 2024 were included in the continuous observation period.

According to the study design characteristics, the intervention will be performed on the control group after the randomized controlled trial phase and the sustainability of the initial intervention group after 3 months will be assessed. The intervention group started in January 2024, implemented the validated intervention protocol and quality promotion implementation strategy, and entered the second phase three months later (April 2024), and the control group became the second intervention group after the intervention in April 2024. In Phase I (the randomized controlled trial phase, January 2024 to March 2024), the effect of the intervention and the improvement strategy was examined by comparing the change in BSI at baseline between the two groups. The control group started the intervention (January 2024) and began reporting bloodstream infection data. In the second phase (April 2024 to June 2024), both groups received the intervention and were followed up until September 2024. Therefore, it is possible to observe the first intervention group for 9 months and also to verify whether the results of the second intervention group (the phase I control group) can be replicated.

Control group: According to hospital catheterization, maintenance and central venous catheter extraction routine care.

Intervention group: On the basis of routine care, the "evidence-based intervention Program for the Prevention of Catheter Related bloodstream infection (CRBSI) in ICU patients" was implemented for intervention.

Primary outcome: incidence of CRBSI, ratio of CRBSI incidence (quarterly comparison) Secondary outcome ：length of stay in ICU, BSI-related mortality in ICU, hospitalization cost in ICU, knowledge and practice score of adherence to evidence-based sensory control in ICU, adherence to evidence-based practice of central venous catheter placement, maintenance and extubation.

ELIGIBILITY:
Inclusion Criteria:

* ICU stay over 48 hours
* CVC was placed for more than 24 hours

Exclusion Criteria:

* Pregnant patients
* Patients with a history of CRBSI infection
* Patients with central venous catheterization were brought in from other hospitals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8050 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of CRBSI | 1year
CRBSI incidence ratio | 1 year
  Ratio of CRBSI incidence per quarter (IRR)

SECONDARY OUTCOMES:
Length of ICU stay | 1 year
  Length of ICU stay
Related Mortality | 1 year
  ICU CRBSI-related mortality
ICU hospitalization cost | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yan Hu, Study Chair — School of Nursing, Fudan University; Center for Evidence-based Nursing, Fudan University; YuXia Zhang, Study Director — Department of Nursing, Zhongshan Hospital Affiliated to Fudan University; Ying Gu, Study Director — Center for Evidence-based Nursing, Fudan University
Locations (1):
- ZhongShan Hospital Affilicated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The research institute shares research data and results according to the plan. The materials and data involved in the study are for the research group only. The final interpretation belongs to the research group
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The materials and data involved in the study are available for five years from the start of the study to the end of the study, and the results of the study are agreed to be used for the study itself.
Access Criteria: Provide access to the head of each research branch or PI

REFERENCES:
- [Result] Peng S, Lu Y. Clinical epidemiology of central venous catheter-related bloodstream infections in an intensive care unit in China. J Crit Care. 2013 Jun;28(3):277-83. doi: 10.1016/j.jcrc.2012.09.007. Epub 2012 Dec 21. PMID 23265289
- [Result] Lindgren S, Pikwer A, Ricksten SE, Akeson J. Survey of central venous catheterisation practice in Sweden. Acta Anaesthesiol Scand. 2013 Nov;57(10):1237-44. doi: 10.1111/aas.12190. Epub 2013 Sep 16. PMID 24102163
- [Result] Govindan S, Jobe A, O'Malley ME, Flanders SA, Chopra V. To PICC or not to PICC? A cross-sectional survey of vascular access practices in the ICU. J Crit Care. 2021 Jun;63:98-103. doi: 10.1016/j.jcrc.2021.02.004. Epub 2021 Feb 20. PMID 33652363
- [Result] Parienti JJ, Mongardon N, Megarbane B, Mira JP, Kalfon P, Gros A, Marque S, Thuong M, Pottier V, Ramakers M, Savary B, Seguin A, Valette X, Terzi N, Sauneuf B, Cattoir V, Mermel LA, du Cheyron D; 3SITES Study Group. Intravascular Complications of Central Venous Catheterization by Insertion Site. N Engl J Med. 2015 Sep 24;373(13):1220-9. doi: 10.1056/NEJMoa1500964. PMID 26398070
- [Result] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee (HICPAC). Guidelines for the prevention of intravascular catheter-related infections. Clin Infect Dis. 2011 May;52(9):e162-93. doi: 10.1093/cid/cir257. Epub 2011 Apr 1. No abstract available. PMID 21460264
- [Result] Rosenthal VD, Maki DG, Mehta Y, Leblebicioglu H, Memish ZA, Al-Mousa HH, Balkhy H, Hu B, Alvarez-Moreno C, Medeiros EA, Apisarnthanarak A, Raka L, Cuellar LE, Ahmed A, Navoa-Ng JA, El-Kholy AA, Kanj SS, Bat-Erdene I, Duszynska W, Van Truong N, Pazmino LN, See-Lum LC, Fernandez-Hidalgo R, Di-Silvestre G, Zand F, Hlinkova S, Belskiy V, Al-Rahma H, Luque-Torres MT, Bayraktar N, Mitrev Z, Gurskis V, Fisher D, Abu-Khader IB, Berechid K, Rodriguez-Sanchez A, Horhat FG, Requejo-Pino O, Hadjieva N, Ben-Jaballah N, Garcia-Mayorca E, Kushner-Davalos L, Pasic S, Pedrozo-Ortiz LE, Apostolopoulou E, Mejia N, Gamar-Elanbya MO, Jayatilleke K, de Lourdes-Duenas M, Aguirre-Avalos G; International Nosocomial Infection Control Consortium. International Nosocomial Infection Control Consortium (INICC) report, data summary of 43 countries for 2007-2012. Device-associated module. Am J Infect Control. 2014 Sep;42(9):942-56. doi: 10.1016/j.ajic.2014.05.029. PMID 25179325
- [Result] Granger BB. Science of Improvement Versus Science of Implementation: Integrating Both Into Clinical Inquiry. AACN Adv Crit Care. 2018 Summer;29(2):208-212. doi: 10.4037/aacnacc2018757. No abstract available. PMID 29875118
- [Result] Koczwara B, Stover AM, Davies L, Davis MM, Fleisher L, Ramanadhan S, Schroeck FR, Zullig LL, Chambers DA, Proctor E. Harnessing the Synergy Between Improvement Science and Implementation Science in Cancer: A Call to Action. J Oncol Pract. 2018 Jun;14(6):335-340. doi: 10.1200/JOP.17.00083. Epub 2018 May 14. No abstract available. PMID 29750579
- [Result] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537
- [Result] Berenholtz SM, Lubomski LH, Weeks K, Goeschel CA, Marsteller JA, Pham JC, Sawyer MD, Thompson DA, Winters BD, Cosgrove SE, Yang T, Louis TA, Meyer Lucas B, George CT, Watson SR, Albert-Lesher MI, St Andre JR, Combes JR, Bohr D, Hines SC, Battles JB, Pronovost PJ; On the CUSP: Stop BSI program. Eliminating central line-associated bloodstream infections: a national patient safety imperative. Infect Control Hosp Epidemiol. 2014 Jan;35(1):56-62. doi: 10.1086/674384. Epub 2013 Nov 26. PMID 24334799
- [Result] Marsteller JA, Sexton JB, Hsu YJ, Hsiao CJ, Holzmueller CG, Pronovost PJ, Thompson DA. A multicenter, phased, cluster-randomized controlled trial to reduce central line-associated bloodstream infections in intensive care units*. Crit Care Med. 2012 Nov;40(11):2933-9. doi: 10.1097/CCM.0b013e31825fd4d8. PMID 22890251
- [Result] Blot K, Bergs J, Vogelaers D, Blot S, Vandijck D. Prevention of central line-associated bloodstream infections through quality improvement interventions: a systematic review and meta-analysis. Clin Infect Dis. 2014 Jul 1;59(1):96-105. doi: 10.1093/cid/ciu239. Epub 2014 Apr 9. PMID 24723276
- [Result] Gorski LA. The 2016 Infusion Therapy Standards of Practice. Home Healthc Now. 2017 Jan;35(1):10-18. doi: 10.1097/NHH.0000000000000481. PMID 27922994
- [Result] Septimus EJ. Society for Healthcare Epidemiology of America Compendium updates 2022. Curr Opin Infect Dis. 2023 Aug 1;36(4):263-269. doi: 10.1097/QCO.0000000000000926. Epub 2023 Jun 2. PMID 37260268
- [Derived] Zhou T, Li C, Wang Z, Yang M, He X, Hu Y. Evidence-Based Practice in Maintenance of Central Venous Catheters Among Intensive Care Unit Nurses: A Cross-Sectional Multi-Center Study. J Clin Nurs. 2025 Oct;34(10):4351-4365. doi: 10.1111/jocn.17692. Epub 2025 Mar 24. PMID 40125637